CLINICAL TRIAL: NCT01797406
Title: Water Injection Colonoscopy vs Air Insufflation Colonoscopy in Experienced Endoscopists
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: WIC-003
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Colon Disease;; Rectal Disease;
MeSH Terms: conditions — Colonic Diseases; Rectal Diseases | interventions — Water

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Air insufflation colonoscopy (Active Comparator): Air insufflation colonoscopy is the conventional colonoscopy,which is inflating air to help searching the bowel cavity while advancing the colonoscope until reaching the cecum.All the patients were examined without sedation during the whole procedure.
  Interventions: Other: Air insufflation
- Water injection colonoscopy (Experimental): Water injection colonoscopy : Cut off air inflating before examination. Water was injected through the working channel to follow the intestinal cavity until reaching the caecum .All the patients were examined without sedation during the whole procedure.
  Interventions: Other: Water injection

INTERVENTIONS:
Other: Air insufflation — Air is inflated into the bowel to help searching the cavity while advancing the colonoscope until reaching the cecum
  Arms: Air insufflation colonoscopy
Other: Water injection — Water was injected through the working channel instead of air to follow the intestinal cavity until reaching the caecum .
  Arms: Water injection colonoscopy

SUMMARY:
Water injection colonoscopy has been a generally accepted method in training the beginners of colonoscopy for its low pain and less cecal intubation time, the investigators would conduct this study to investigate advantages of this method for experienced endoscopists.

DETAILED DESCRIPTION:
Up to now, many studies has showed that compared with air insufflation colonoscopy, water-related colonoscopy could shorten the cecal intubation time and relieve the pain of the patients,especially for training the beginners，the effect was notable, but the present researches on water assisted technique has still been confined to following aspects:1.Water infusing was based on air insufflation; predetermined amount of water was infused ,and water was infused while passing through certain segment of the bowel(such as the left half of colon) ; 2.When training the first-learners, certain dose of sedatives or analgesics was injected; 3.The patients recruited were less. Colonoscopies in this study would be performed by experienced endoscopists of air insufflation colonoscopy, water would be injected completely instead of air insufflation while advancing the colonoscope, the amount of the water infused would not be predetermined but vary from individuals, and all the patients would be examined without any sedatives or analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnostic colonoscopy;
* Subjets able to provide informed consent

Exclusion Criteria:

* Prior partial or complete colectomy;
* Patients who decline to participate;
* Patients with poor bowel preparation;
* Contraindications of the colonoscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
The success rate of the cecal intubation | This will be calculated after the completion of the whole trial,which is about 2 months

SECONDARY OUTCOMES:
The cecal intubation time(min); | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length
The time to reach the splenic flexure(min) | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length
VAS abdominal pain score | Data collected usually within 10minutes post procedure
The frequency of the colonoscope shortening maneuver while advancing the colonoscope | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length.
Length of colonoscope at time of cecal intubation(cm) | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length.
Volume of water used during water colonoscopy(ml) | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length.
General data of the patients recruited-age | Data collected usually within 10minutes post procedure .
General data of the patients recruited-gender | Data collected usually within 10minutes post procedure .
General data of the patients recruited-BMI | Data collected usually within 10minutes post procedure .
General data of the patients recruited-abdominal or pelvic surgery history | Data collected usually within 10minutes post procedure .
General data of the patients recruited-bowel preparation | Data collected usually within 10minutes post procedure .
The McGill pain evaluation of the abdominal pain | Data collected usually within 10minutes post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Youlin Yang, M.D., Principal Investigator — The Gastroenterology Department of the 1st Affiliated Hospital of Harbin Medical University
Locations (1):
- The Gastroenterology Department of the 1st Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China